CLINICAL TRIAL: NCT03252964
Title: Empowering Medicare Patients to Self-Manage Their Type 2 Diabetes Using Continuous Glucose Monitoring (CGM) - Investigational Device Pilot
Brief Title: Continuous Glucose Monitors to Regulate Glucose Levels in Type 2 Diabetics
Acronym: CGM_IRB2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Savvysherpa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00021722
Record Dates: First submitted 2017-08-09; First posted 2017-08-17 (Actual); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Fitness Trackers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Diabetes Management Educational Program (Experimental): Subjects receive a CGM and activity tracker as part of a educational program to help manage their glucose levels.
  Interventions: Device: Continuous Glucose Monitor (CGM); Device: Activity Tracker; Behavioral: Coaching

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — Subjects will use a CGM to develop an understanding of how their behaviors influence their glucose levels.
  Other Names: Dexcom Investigational Use Only (IUO) Device
Device: Activity Tracker — Subjects will use the activity tracker, in combination with a continuous glucose monitor (CGM), to develop an understanding of how their activity levels affect their glucose levels.
  Other Names: Fitbit Charge 2
Behavioral: Coaching — Coaches will help subjects understand the readings from the CGMs and how they are affected by diet choices, use of diabetes medications, etc. Coaches and subjects will have weekly conversations about CGM data and behaviors that affect CGM readings. Coaching will occur via telephone, text messaging, and automated text messaging.

SUMMARY:
This study allows Type 2 diabetics to receive feedback from a continuous glucose monitor (CGM) as part of an educational program designed to help them better manage their glucose levels. Subjects will also wear an activity tracker to monitor their activity and observe its effect on their glucose levels. The educational program will involve calls from coaches to check subjects' progress and answer questions.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with type 2 diabetes
* Currently take a DPP4 inhibitor, SGLT2 inhibitor, GLP-1 agonist, and/or basal insulin
* Be able to read and understand English
* Have access to a telephone
* Have a Medicare health plan

Exclusion Criteria:

* Pregnant
* Blind
* Deaf
* Currently receiving chemotherapy or radiation therapy to treat cancer
* Addicted to any drugs (including alcohol, painkillers, hallucinogens, or others)
* Critically ill
* Diagnosed with or experiencing:

  * Kidney disease stages 4 and 5
  * End stage renal disease
  * Severe liver disease
  * Dementia
  * Schizophrenia
  * Bipolar disorder
  * Autism
  * An intellectual or learning disability
  * Arrhythmias other than atrial fibrillation
  * Congestive heart failure
* Has had a:

  * Myocardial infarction within the last 6 months
  * Stroke within the last 6 months
  * Stroke that resulted in significant disability (e.g., unable to write clearly or walk)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rogelio Machuca, MD Family Medicine, PLLC, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 364 candidates were contacted. Of those, 52 enrolled.
Period: Overall Study
Arm/Group | Diabetes Management Educational Program
Started | 52
Completed | 20
Not Completed | 32

BASELINE CHARACTERISTICS:
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Program Enrollment Rate (%)
Description: (Number of patients who signed a consent form)/(Number of patients invited to enroll)
Time Frame: up to three months
Population: 52 participants enrolled in the study. Hence, 52 participants analyzed. However, enrollment rate is the number of participants enrolled (52) divided by the number of candidates contacted (364). This explains why the Overall Number of Participants Analyzed is greater than the number Started in the Participant Flow.
Measure: Number; unit: Percentage of participants
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 364
Percentage of participants | 14

2. Primary Outcome: Program Completion Rate (%)
Description: (Number of patients who complete 49 days of CGM use) / (Number of patients who signed the consent form)
Time Frame: up to six months
Measure: Number; unit: Percentage of participants
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 52
Percentage of participants | 38

3. Secondary Outcome: Change in A1c Measurement (%)
Description: (Final A1c measure)-(Initial A1c measure)
Time Frame: Day 0 and Day 180
Population: Lack of study resources to collect sufficient information on this variable.
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 0

4. Secondary Outcome: Weekly Average of Estimated Glucose Values (EGV) (Average)
Description: (Sum of EGV for one week)/(Total number of EGV)
Time Frame: up to six months
Population: Lack of study resources to collect sufficient information on this variable.
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Medication Dosage (mg/Day; U/Day)
Description: (dosage of Rx on Day 180)-(dosage of Rx on Day 0)
Time Frame: up to six months
Population: Lack of study resources to collect adequate information on this variable.
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 0

6. Secondary Outcome: Average Age of Participants Who Start Trial (Yrs)
Description: (Sum of ages of all enrollees)/(Total number of enrollees)
Time Frame: up to three months
Population: Lack of study resources to collect adequate information on this variable.
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 0

7. Secondary Outcome: Average Age of Participants Who Complete Trial (Yrs)
Description: (Sum of age of patients who complete)/(Total number who complete)
Time Frame: up to six months
Population: Lack of study resources to collect sufficient data on outcome variable.
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 0

8. Secondary Outcome: Race of Participants Who Start the Trial (n)
Description: Sum of American Indian or Alaska Native, Sum of Asian, Sum of Black or African American, Sum of Native Hawaiian or Other Pacific Islander, Sum of White
Time Frame: up to three months
Population: Lack of study resources to collect sufficient data on outcome variable.
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 0

9. Secondary Outcome: Ethnicity of Participants Who Start the Trial (n)
Description: Sum of Hispanic or Latino and Sum of Not Hispanic or Latino
Time Frame: up to three months
Population: Lack of study resources to collect sufficient data on outcome variable.
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 0

10. Secondary Outcome: Texting With Coaches (Daily Average of Text Messages)
Description: (Sum of all text messages)/(Total number of days)
Time Frame: up to six months
Population: Lack of study resources to collect sufficient data on outcome variable.
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 0

11. Secondary Outcome: Coaching Participation Rate
Description: (Sum of weekly coaching calls completed)/(Total number of weeks)
Time Frame: up to six months
Population: Lack of study resources to collect sufficient data on outcome variable.
Arm/Group | Diabetes Management Educational Program
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 8 months
Description: AE and SAE were monitored in three ways:
  * Participants were instructed to call the study doctor's clinical research coordinator (CRC) to report all AE and SAE related to the study devices.
  * Study coaches listened for any reports of AE or SAE in their communications with participants and connected reporting patients with the CRC.
  * Reports of AE or SAE received by Dexcom's Customer Care and Technical Support representatives were documented and reported to the Sponsor and CRC.
Arm/Group | Diabetes Management Educational Program
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 2/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diabetes Management Educational Program (N=52)
Bleeding (Skin and subcutaneous tissue disorders) | 1 — Bleeding at CGM sensor insertion site.
Pain (Skin and subcutaneous tissue disorders) | 1 — Pain at CGM sensor insertion site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT03252964/Prot_000.pdf
  • Informed Consent Form (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03252964/ICF_001.pdf